CLINICAL TRIAL: NCT01622764
Title: 89Zr-RO5323441 PET Imaging in Patients With Recurrent Glioblastoma Treated With Bevacizumab
Brief Title: 89Zr-RO5323441 PET Imaging in Glioblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding from the sponsor
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BP28015; 2011-004974-27 (EudraCT Number)
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Glioblastoma
Keywords: RO5323441; bevacizumab; PET imaging; recurrent glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Molecular Imaging; TB-403

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Molecular imaging with 89Zr-RO5323441 (Experimental)
  Interventions: Radiation: Molecular imaging with 89Zr-RO5323441

INTERVENTIONS:
Radiation: Molecular imaging with 89Zr-RO5323441 — Bevacizumab at a dose of 10 mg/kg body weight i.v. in 90 min on day 1 will be given every 2 weeks in cycles of 6 weeks, until documented disease progression, unacceptable toxicity, patient refusal or patient's best interest. 89Zr-RO5323441 will be administered i.v. at a tracer dose of 5 mg (37 MBq) on day -3 and on day 11 of cycle 1 of bevacizumab treatment. Four PET scans will be performed (2 brain only PET scans and 2 whole body PET scans). Brain only PET scans will be performed 2 hours after each 89Zr-RO5323441 administration on day -3 and day 11. Whole body PET scans will be performed 4 days after each 89Zr-RO5323441 administration (before dosing with bevacizumab on day 1 and day 15).
  Other Names: TB403

SUMMARY:
The research the investigators propose is a molecular imaging study of RO5323441, an antibody against placental growth factor (PlGF) in patients with recurrent GBM treated with bevacizumab, a drug against vascular endothelial growth factor (VEGF). Both VEGF and PlGF are molecules involved in tumor growth since they enable the development of tumor vasculature, thus delivery of oxygen and nutrients to the tumor. The treatment will consist of bevacizumab (i.v.) given every 2 weeks, until the patient has clinical benefit (no disease progression) or unacceptable toxicity. Meanwhile, patients will receive and injection of low protein-dose radiolabeled RO5323441 (89Zr-RO5323441) on day -3 and 11 of the first bevacizumab treatment cycle. Brain-only 89Zr-RO5323441 positron emission tomography (PET) will be performed at 2 hours after each injection of 89Zr-RO5323441 on day -3 and 11. Whole body 89Zr-RO5323441 PET will be performed on day 1 and 15, before and after the first treatment with bevacizumab. The main purpose of this trial is to determine how much of RO5323441 actually gets into the recurrent GBM lesions, since for a drug to be active, it has to be able to reach cancer cells. As second aims, RO5323441 accumulation in normal, non-tumor organs, will be assessed, as well as how bevacizumab influences RO5323441 penetration into tumor lesions (to answer the question of combined bevacizumab + RO5323441 treatment in GBM) or RO5323441 biodistribution in non-tumor organs.

DETAILED DESCRIPTION:
Rationale: Glioblastomas (GBM) account for 70% of all gliomas (80% of all malignant brain and CNS tumors) and remain the most aggressive sub-type of glioma, with a particularly poor prognosis. Surgery aimed to complete resection is the first therapeutic modality, however, the infiltrative nature of the disease makes a complete resection nearly impossible. In a randomized, phase III EORTC-NCIC trial, overall survival in newly diagnosed glioblastoma patients treated with concomitant temozolomide and radiotherapy followed by 6 cycles of temozolomide was 27.2% (95% CI 22.2-32.5) at 2 years, 16.0% (12.0-20.6) at 3 years, 12.1% (8.5-16.4) at 4 years, and 9.8% (6.4-14.0) at 5 years, treatment which is now standard of care. Almost all GBM patients experience relapse and there is no one generally agreed standard of care in recurrent GBM. Vascular endothelial growth factor-A (VEGF-A), a central regulator of physiological and pathological angiogenesis, is considered to play a major angiogenic role in GBM. Bevacizumab, a humanized monoclonal antibody against VEGF-A, showed a 28%RR,a 43% 6-month PFS and provided a consistent clinical benefit in terms of both delayed progression and increased median overall survival over historical controls. This benefit is limited however, with the tumor eventually evading treatment by for example compensatory upregulation of angiogenic factors like placental growth factor (PlGF). Therefore, targeting PlGF could be a new strategy of tumor angiogenesis inhibition, complementary to VEGF(R) inhibition. In preclinical setting, inhibiting PlGF has shown to inhibit growth and metastasis of various tumors. Humanized monoclonal PlGF antibody RO5323441 was evaluated in phase I trials in healthy volunteers and in cancer patients; no Dose Limiting Toxicity (DLT) was found, thus no Maximum Tolerated Dose (MTD) defined. Stable disease was observed in 6/23 patients on different dose levels. A phase I/II study of bevacizumab in combination with RO5323441 is currently ongoing in patients with recurrent GBM (NCT01308684). However, the amount of RO5323441 to reach the recurrent GBM, and how this is affected by bevacizumab treatment, are yet unknown. This can be determined by repetitive measurement of RO5323441 tumor uptake with 89Zr-RO5323441 PET.

Objectives: The objectives of this study are to assess the penetration of RO532441 into recurrent GBM by 89Zr-RO5323441 PET imaging and to quantify its uptake, to visualize and quantify 89Zr-RO5323441 non-tumor organ distribution, and to measure the effect of bevacizumab treatment on 89Zr-RO5323441 uptake in recurrent GBM.

Study design: This is a single center, investigator driven, 89Zr-RO5323441 PET imaging and bio-distribution study in patients with recurrent GBM treated with bevacizumab. Bevacizumab at a dose of 10 mg/kg body weight i.v. in 90 min on day 1 is given every 2 weeks in cycles of 6 weeks. The treatment with bevacizumab will continue until documented disease progression, unacceptable toxicity, patient refusal or patient's best interest. 89Zr-RO5323441 will be administered i.v. at a tracer dose of 5 mg (37 MBq) on day -3 and on day 11 of cycle 1 of bevacizumab treatment. Four PET scans will be performed (2 brain only PET scans and 2 whole body PET scans). Brain only PET scans will be performed 2 hours after each 89Zr-RO5323441 administration on day -3 and day 11, and will take 10 minutes/ scan. Whole body PET scans will be performed 4 days after each 89Zr-RO5323441 administration (before dosing with bevacizumab on day 1 and day 15), and will take 50 minutes/ scan. 89Zr-RO5323441 uptake values in recurrent GBM lesions at baseline and day 15 will be compared to assess bevacizumab effect on tracer tumor uptake. The purpose of the two early brain-only PET scans after each 89Zr-RO5323441 injection is to identify whether changes in 89Zr-RO5323441 uptake in recurrent GBM lesions following treatment with bevacizumab can be solely attributed to an effect on blood volume/ vascular permeability, or rather indicate a possible modulation of placental growth factor (PlGF) level in the tumor tissue. The rationale for the whole body 89Zr-RO5323441 PET scans is to assess 89Zr-RO5323441 non-tumor organs distribution at baseline, as well as to evaluate the influence bevacizumab treatment could exert on 89Zr-RO5323441 non-tumor organs uptake. For 89Zr-RO5323441 pharmacokinetics, blood samples will be taken 1 hour after 89Zr-RO5323441 tracer injection on d-3 and d11, respectively together with the blood samples for hematology on d1 and d15 during the 1st cycle of bevacizumab treatment. The rationale for this is that performing both the 89Zr-RO5323441 PET scan data quantification and the assessment of the tracer's blood pharmacokinetics would enable us to better understand the specificity of 89Zr-RO5323441 uptake in recurrent GBM lesions. Patients will be assessed for bevacizumab treatment response by brain MRI every 6 weeks (i.e. every cycle) in the first 6 month and every 12 weeks thereafter, until documented progression using the updated RANO criteria. Treatment and tracer injection related side effects will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE; version 4.0) for toxicity and adverse event reporting.

Main study parameters/ endpoints: 89Zr-RO5323441 tumor uptake and organ distribution will be scored visually and quantitatively. Standardized uptake value (SUV) and relative uptake value (RUV) will be determined and compared in the recurrent GBM lesions and in relevant tissues at baseline and day 15.

Nature and extent of the burden and risk associated with participation, benefit and group relatedness: Bevacizumab is registered in The Netherlands for use in metastasized colon and breast cancer, in lung cancer and in advanced renal cell carcinoma and has already been tested in GBM clinical trials. Bevacizumab is expected to have clinical benefit for patients enrolled in this study and similar safety profile compared to the other indications. RO5323441 monotherapy was well tolerated in patients with advanced malignant diseases. In this study, one patient will receive a low total protein dose of 10 mg RO5323441 (2X5mg) in the tracer and it is expected that RO5323441 will not enhance bevacizumab related side effects. The total radiation dose of 89Zr-RO5323441 for a patient participating in this study would be 36 mSv for women and 30 mSv for men. According to the investigators this radiation burden is justifiable in this patient group by the information that can be obtained in this study. Risk: exposure to 89Zr-RO5323441 PET scan-related radiation, possibility of allergic reaction to the protein in the tracer, possible side-effects of bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Age more or at least equal to 18 years
* WHO Performance Status between 0 and 2
* Histologically proven glioblastoma multiforme at recurrence, including patients with anaplastic oligoastrocytomas with necrosis
* Patients treated with one line of systemic treatment (combined treatment with temozolomide and RT followed by 6 cycles of temozolomide is considered as one line of systemic treatment)
* No prior treatment with bevacizumab or other PlGF,VEGF,VEGF-R targeted agents, cilengitide or enzastaurin
* No radiotherapy within 4 weeks prior to the diagnosis of progression
* No chemotherapy within 4 weeks prior to study enrollment
* Adequate bone marrow function
* Adequate liver function
* Adequate renal function
* Women of reproductive potential, female patients within one year of entering the menopause as well as males must agree to use an effective non-hormonal method of contraception during the treatment period and for at least 6 months after the last dose of bevacizumab
* Written informed consent

Exclusion Criteria:

* Invasive procedures (major surgical procedure, open biopsy or significant traumatic injury) within 28 days prior to start study treatment, or anticipation of the need for major surgery during the course of the study treatment. Placement of a vascular access device is not considered as a major surgical procedure if performed more than 24 hours prior to bevacizumab administration.
* Arterial or venous thrombosis less or equal than 6 months prior to study registration
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History of myocardial infarction (less or equal than 6 months prior to inclusion), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring digoxin treatment
* Uncontrolled hypertension defined by a systolic blood pressure (BP) more than 140 mm Hg and or diastolic pressure more than 100 mm Hg, with or without anti-hypertensive medication. Patients with initial blood pressure elevation are eligible if initiation or adjustment of anti-hypertensive medication lowers pressure to meet the entry criteria
* History or evidence of inherited bleeding diathesis or coagulopathy with risk of bleeding
* Current or recent (within 10 days of first dose of bevacizumab) use of aspirin more than 325 mg per day) or other NSAID with anti-platelet activity or treatment with dipyramidole, ticlopidine, clopidogrel and cilostazol
* Use of therapeutic-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic (as opposed to prophylactic) purposes
* Clinically serious (as judged by the investigator) non-healing wounds, active skin ulcers or incompletely healed bone fracture
* Evidence of any active infection requiring hospitalization or antibiotics, within 2 weeks prior to day 1 of cycle 1
* Current or recent (within 4 weeks of enrollment) treatment with another investigational drug or participation in another investigational study
* Known hypersensitivity to any part of the bevacizumab formulation
* Hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibody
* Other diseases, interfering with the follow-up
* Geographical, psychological or other non-medical conditions interfering with follow-up
* Pregnant or lactating females (serum pregnancy test to be assessed before entry in the trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Assess the penetration of RO5323441 into recurrent GBM by 89Zr-RO5323441 PET imaging and to quantify its uptake | Patients will be assessed up to 19 days after the first 89Zr-RO5323441 tracer injection (D-3)
  Calculations of specific 89Zr-RO5323441 uptake in recurrent GBM lesions will be determined for all patients who underwent tracer injection(s) and 89Zr-RO5323441 PET. 89Zr-RO5323441 tumor uptake will be scored visually and quantitatively. The visual analysis of the PET scans will be performed by a qualified nuclear medicine physician. Quantification of 89Zr-RO5323441 uptake will be performed using AMIDE software (Stanford University, Palo Alto, CA). Standardized uptake value (SUV) and relative uptake value (RUV)of 89Zr-RO5323441 will be determined.

SECONDARY OUTCOMES:
Visualize and quantify 89Zr-RO5323441 non-tumor organ distribution | Patients will be assessed up to 19 days after the first 89Zr-RO5323441 tracer injection (D-3)
  89Zr-RO5323441 non-tumor organs biodistribution will be determined for all patients who underwent tracer injection(s)and 89Zr-RO5323441 PET. 89Zr-RO5323441 non-tumor organs biodistribution will be scored visually and quantitatively. The visual analysis of the PET scans will be performed by a qualified nuclear medicine physician. Quantification of 89Zr-RO5323441 biodistribution in non-tumor organs will be performed using AMIDE software (Stanford University, Palo Alto, CA).
Assess the effect of bevacizumab treatment on 89Zr-RO5323441 uptake in recurrent GBM lesions | Patients will be assessed up to 19 days after the first 89Zr-RO5323441 tracer injection, which also corresponds to the second bevacizumab dose administered
  89Zr-RO5323441 uptake values in recurrent GBM lesions at baseline and day 15 will be compared to assess bevacizumab effect on tracer tumor uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Annemiek M. Walenkamp, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands